CLINICAL TRIAL: NCT05157269
Title: Phase 3, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate Efficacy and Safety of Nitazoxanide in the Treatment of Mild COVID-19 in Subjects Not at High Risk of Severe Illness
Brief Title: Trial to Evaluate Nitazoxanide for Treatment of Mild COVID-19 in Subjects Not at High Risk of Severe Illness
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Romark Laboratories L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RM08-3011
Record Dates: First submitted 2021-12-10; First posted 2021-12-14 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: COVID-19
Keywords: SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — nitazoxanide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nitazoxanide (Active Comparator): Nitazoxanide 300 mg extended release tablets
  Interventions: Drug: Nitazoxanide; Dietary Supplement: Vitamin Super-B Complex
- Placebo (Placebo Comparator): Placebo tablets
  Interventions: Drug: Placebo; Dietary Supplement: Vitamin Super-B Complex

INTERVENTIONS:
Drug: Nitazoxanide — Two NTZ 300 mg extended release tablets administered orally with food twice daily for 5 days
  Other Names: NTZ; NT-300
  Arms: Nitazoxanide
Drug: Placebo — Two matching placebo tablets administered orally twice daily for 5 days
  Arms: Placebo
Dietary Supplement: Vitamin Super-B Complex — Vitamin Super-B Complex administered orally with food twice daily for 5 days to maintain the blind

SUMMARY:
The purpose of this study is to determine whether nitazoxanide (NTZ) is safe and effective for treatment of mild COVID-19 illness. Adults and adolescent participants will be followed for approximately 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 12 years of age
* Positive test for SARS-CoV-2 by RT-PCR or validated rapid antigen test within 72 hours prior to enrollment in the trial (positive sample must be collected within 72 hours prior to enrollment).
* Presence of clinical signs and/or symptoms consistent with worsening or stable mild COVID-19 (one of the following is required):

  1. Presence of at least two respiratory symptom domains (head, throat, nose, chest, cough) with a score of ≥2 as determined by Screening FLU-PRO AND
  2. Patient reported assessment that symptoms are present, the symptoms are not consistent with the subject's usual health, the symptoms interfere with daily activities, and the symptoms have worsened or remained the same relative to the previous day, as confirmed by responses to questions in the Screening FLU-PRO.
* Onset of symptoms no more than 72 hours before enrollment in the trial. Onset of symptoms is defined as the earlier of the first time at which the subject experienced subjective fever or any respiratory symptom (headache/head congestion, throat symptoms, nasal symptoms, chest symptoms, cough).
* Willing and able to provide written informed consent (including assent by legal guardian if under 18 years of age) and comply with the requirements of the protocol, including completion of the subject diary and all protocol procedures.

Exclusion Criteria:

* Persons with any clinical sign or symptoms suggestive of moderate or severe systemic illness with COVID-19, including the following:

  1. shortness of breath at rest,
  2. resting pulse ≥90 beats per minute,
  3. resting respiratory rate ≥20 breaths per minute, or
  4. oxygen saturation ≤ 93% on room air at sea level.
* Persons who have not been fully vaccinated against SARS-CoV-2 and are at high risk of progressing to severe COVID-19 illness due to having one of the following underlying conditions and/or sociodemographic risk factors:

  1. Age ≥ 55 years (with or without comorbidities),
  2. Body mass index (BMI) ≥30 kg/m² if ≥ 18 years of age or BMI ≥85th percentile for age and gender based on CDC growth charts,
  3. Chronic kidney disease,
  4. Diabetes,
  5. Cardiovascular disease (including congenital heart disease) or hypertension,
  6. Chronic lung disease (e.g., chronic obstructive pulmonary disease, moderate-to-severe asthma, interstitial lung disease, cystic fibrosis, pulmonary hypertension),
  7. Sickle cell disease,
  8. Neurodevelopmental disorders or other conditions that confer medical complexity.
* Subjects with immunosuppressive disease or receiving immunosuppressive treatment regardless of SARS-CoV-2 vaccination status.
* Subjects with active respiratory allergies or subjects expected to require anti-allergy medications during the study period for respiratory allergies.
* Females of childbearing potential who are either pregnant or sexually active without the use of birth control.
* Subjects residing in the same household with another subject participating in the study.
* Treatment with any investigational drug or vaccine therapy within 30 days prior to screening and willing to avoid them during the course of the study.
* Subjects who have received within the past 90 days or are expected to receive during the study period monoclonal antibody treatment or convalescent COVID-19 plasma for COVID-19.
* Receipt of any dose of NTZ within seven days prior to screening.
* Known sensitivity to NTZ or any of the excipients comprising the study medication.
* Subjects unable to swallow oral tablets or capsules.
* Subjects with known severe heart, lung, neurological or other systemic disease that the Investigator believes could preclude safe participation.
* Subjects likely or expected to require hospitalization unrelated to COVID-19 during the study period.
* Subjects taking medications considered to be major CYP2C8 substrates.
* Subjects who, in the judgment of the Investigator, will be unlikely to comply with the requirements of this protocol including completion of the subject diary.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Time to sustained COVID-19 Recovery | Day 1 through Day 21

OTHER OUTCOMES:
Time to return to usual health | Day 1 through Day 21
Proportion of participants progressing to severe COVID-19 illness or death by any cause | Day 1 through Day 28
Change in cytokine levels | Day 1 through Day 4